CLINICAL TRIAL: NCT00407186
Title: A Multicenter Randomized Phase III Trial of Neo-adjuvant Chemotherapy Followed by Surgery and Chemotherapy or by Surgery and Chemoradiotherapy in Resectable Gastric Cancer (CRITICS Study)
Brief Title: Randomized Phase III Trial of Adjuvant Chemotherapy or Chemoradiotherapy in Resectable Gastric Cancer (CRITICS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dutch Colorectal Cancer Group (Other)
Collaborators: The Netherlands Cancer Institute (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRITICS
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Gastric Cancer
Keywords: CRITICS; gastric cancer; surgery; adjuvant; chemotherapy; chemoradiotherapy; capecitabine; cisplatin; epirubicin
MeSH Terms: conditions — Stomach Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1chemoradiotherapy (Experimental): 5 weeksadjuvant treatment; radiotherapy and concomitant chemotherapy with cisplatin and capecitabine.
  Interventions: Drug: cisplatin+capecitabine; Radiation: radiotherapy
- 2chemotherapy (Active Comparator): 3 adjuvant courses epirubicin, cisplatin, capecitabine.
  Interventions: Drug: epirubicin+cisplatin+capecitabine

INTERVENTIONS:
Drug: cisplatin+capecitabine — cisplatin 20 mg/m2 (i.v., q 1 w, 5 weeks), capecitabine 575 mg/m2 (b.i.d., oral, on radiotherapy days.
  Arms: 1chemoradiotherapy
Radiation: radiotherapy — 45 Gy in 25 fracions (5 days/week)
  Arms: 1chemoradiotherapy
Drug: epirubicin+cisplatin+capecitabine — 3 courses q 3 w: epirubicin 50 mg/m2 (i.v., day 1), cisplatin 60 mg/m2 (i.v., day 1), capecitabine 1000 mg/m2 (b.i.d., oral, day 1-14)
  Arms: 2chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of combined chemotherapy and radiotherapy (in comparison to chemotherapy alone) as adjuvant treatment after surgery for gastric cancer. Prior to surgery all patients will receive neo-adjuvant chemotherapy as well.

DETAILED DESCRIPTION:
The mainstay of curative treatment of gastric cancer is radical surgical dissection. Because most patients in the Western world present with advanced stages long term survival is found in about 25%, with local recurrences as part of treatment failure in up to 80% of cases. Studies examining the role of more extended lymph node dissections (D1 vs. D2), adjuvant radiotherapy or adjuvant chemotherapy did not result in a clinical relevant improvement of survival. In 2001 results of a South West Oncology group (SWOG) trial that randomized between surgery and surgery with chemoradiotherapy were published. This trial, that was hampered by suboptimal surgery (less than D1 in majority of patients) and radiotherapy (2D radiotherapy; 35% protocol deviations) showed an absolute increase in median survival of 9 months. More recently results of the MAGIC study, which randomized between surgery and surgery plus 6 perioperative courses of ECF chemotherapy, were presented. This regimen resulted in an absolute 5-year survival benefit of 13% and in a 10% higher resectability rate.

This phase III prospectively randomized study investigates whether chemoradiotherapy (45 Gy in 5 weeks with daily cisplatin and capecitabine) after preoperative chemotherapy (3x ECC (epirubicin, cisplatin, capecitabine)) and adequate (D1+) surgery leads to improved survival in comparison with postoperative chemotherapy (3x ECC). Furthermore, toxicity of both treatment regimens will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Ib-IVa (no distant metastases) gastric cancer (histologically proven); tumor bulk in the stomach
* WHO < 2
* Age ≥18 yrs
* Operable gastric cancer
* No prior abdominal radiotherapy or chemotherapy
* Tumornegative laparoscopy when CT suggests peritoneal carcinomatosis
* Start treatment within 10 working days after registration
* Written informed consent

Exclusion Criteria:

* T1N0 disease (endoscopic ultrasound)
* Distant metastases
* Inoperable patients; due to technical surgery-related factors or general condition
* Previous malignancy, except adequately treated non-melanoma skin cancer or in-situ cancer of the cervix uteri.
* Solitary functioning kidney that will be within the radiation field
* Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery
* Uncontrolled (bacterial) infections
* Significant cardiac disorders
* Continuous use of immunosuppressive agents
* Concurrent use of the antiviral agent sorivudine or chemically related analogues
* Hearing loss > CTC grade 1
* Neurotoxicity > CTC grade 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 788 (Actual)
Dates: Start 2007-01-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | study duration

SECONDARY OUTCOMES:
disease-free survival | study duration
toxicity | study duration
health-related quality of life | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Verheij, MD PhD, Principal Investigator — Nederlands Kanker Insituut/Antoni van Leeuwenhoek Ziekenhuis
Locations (1):
- Nederlands Kanker Instituut/Antoni van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands

REFERENCES:
- [Derived] Quaas A, Biesma HD, Wagner AD, Verheij M, van Berge Henegouwen MI, Schoemig-Markiefka B, Pamuk A, Zander T, Siemanowski J, Sikorska K, Egthuijsen JMP, Meershoek-Klein Kranenbarg EM, van de Velde CJH, Buettner R, Alakus H, Cats A, Ylstra B, van Laarhoven HWM, van Grieken NCT. Microsatellite instability and sex differences in resectable gastric cancer - A pooled analysis of three European cohorts. Eur J Cancer. 2022 Sep;173:95-104. doi: 10.1016/j.ejca.2022.06.025. Epub 2022 Jul 18. PMID 35863110
- [Derived] Slagter AE, Vollebergh MA, Caspers IA, van Sandick JW, Sikorska K, Lind P, Nordsmark M, Putter H, Braak JPBM, Meershoek-Klein Kranenbarg E, van de Velde CJH, Jansen EPM, Cats A, van Laarhoven HWM, van Grieken NCT, Verheij M. Prognostic value of tumor markers and ctDNA in patients with resectable gastric cancer receiving perioperative treatment: results from the CRITICS trial. Gastric Cancer. 2022 Mar;25(2):401-410. doi: 10.1007/s10120-021-01258-6. Epub 2021 Oct 29. PMID 34714423
- [Derived] de Steur WO, van Amelsfoort RM, Hartgrink HH, Putter H, Meershoek-Klein Kranenbarg E, van Grieken NCT, van Sandick JW, Claassen YHM, Braak JPBM, Jansen EPM, Sikorska K, van Tinteren H, Walraven I, Lind P, Nordsmark M, van Berge Henegouwen MI, van Laarhoven HWM, Cats A, Verheij M, van de Velde CJH; CRITICS investigators. Adjuvant chemotherapy is superior to chemoradiation after D2 surgery for gastric cancer in the per-protocol analysis of the randomized CRITICS trial. Ann Oncol. 2021 Mar;32(3):360-367. doi: 10.1016/j.annonc.2020.11.004. Epub 2020 Nov 20. PMID 33227408
- [Derived] Slagter AE, Sikorska K, Grootscholten C, van Laarhoven HWM, Lind P, Nordsmark M, Meershoek-Klein Kranenbarg E, van de Velde CJH, van Grieken NCT, van Sandick JW, Jansen EPM, Verheij M, Cats A. Venous thromboembolism during preoperative chemotherapy in the CRITICS gastric cancer trial. Cancer Med. 2020 Sep;9(18):6609-6616. doi: 10.1002/cam4.3118. Epub 2020 Jul 31. PMID 32735752
- [Derived] Slagter AE, Tudela B, van Amelsfoort RM, Sikorska K, van Sandick JW, van de Velde CJH, van Grieken NCT, Lind P, Nordsmark M, Putter H, Hulshof MCCM, van Laarhoven HWM, Grootscholten C, Braak JPBM, Meershoek-Klein Kranenbarg E, Jansen EPM, Cats A, Verheij M. Older versus younger adults with gastric cancer receiving perioperative treatment: Results from the CRITICS trial. Eur J Cancer. 2020 May;130:146-154. doi: 10.1016/j.ejca.2020.02.008. Epub 2020 Mar 21. PMID 32208351
- [Derived] Cats A, Jansen EPM, van Grieken NCT, Sikorska K, Lind P, Nordsmark M, Meershoek-Klein Kranenbarg E, Boot H, Trip AK, Swellengrebel HAM, van Laarhoven HWM, Putter H, van Sandick JW, van Berge Henegouwen MI, Hartgrink HH, van Tinteren H, van de Velde CJH, Verheij M; CRITICS investigators. Chemotherapy versus chemoradiotherapy after surgery and preoperative chemotherapy for resectable gastric cancer (CRITICS): an international, open-label, randomised phase 3 trial. Lancet Oncol. 2018 May;19(5):616-628. doi: 10.1016/S1470-2045(18)30132-3. Epub 2018 Apr 9. PMID 29650363
- [Derived] Dikken JL, van Sandick JW, Maurits Swellengrebel HA, Lind PA, Putter H, Jansen EP, Boot H, van Grieken NC, van de Velde CJ, Verheij M, Cats A. Neo-adjuvant chemotherapy followed by surgery and chemotherapy or by surgery and chemoradiotherapy for patients with resectable gastric cancer (CRITICS). BMC Cancer. 2011 Aug 2;11:329. doi: 10.1186/1471-2407-11-329. PMID 21810227
- [Derived] Jansen EPM, Boot H, Dubbelman R, Verheij M, Cats A. Postoperative chemoradiotherapy in gastric cancer--a phase I-II study of radiotherapy with dose escalation of weekly cisplatin and daily capecitabine chemotherapy. Ann Oncol. 2010 Mar;21(3):530-534. doi: 10.1093/annonc/mdp345. Epub 2009 Aug 18. PMID 19690058
- See also: Dutch Colorectal Cancer Group — http://www.dccg.nl
- See also: Nederlands Kanker Instituut/Antoni van Leeuwenhoek Ziekenhuis (Netherlands Cancer Institute/Antoni van Leeuwenhoek Hospital) — http://www.nki.nl